CLINICAL TRIAL: NCT07174427
Title: Multi-center Study of TBI-1301 (INN: Mipetresgene Autoleucel; Mip-cel) in Patients With NY-ESO-1 Positive Synovial Sarcoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1301-04
Record Dates: First submitted 2025-09-12; First posted 2025-09-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Synovial Sarcomas
Keywords: adoptive cell transfer; NY-ESO-1; T cell receptor; ex vivo gene therapy; synovial sarcoma
MeSH Terms: conditions — Sarcoma, Synovial | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Split dose of 5x10^9 TBI-1301 (Experimental): Split dose of 5x10^9 TBI-1301 will be administered intravenously for 2 days following pre-treatment for 2 days.
  Interventions: Biological: TBI-1301; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: TBI-1301 — Split dose of TBI-1301 is administered intravenously for 2 days following cyclophosphamide/fludarabine pre-treatment.
Drug: Cyclophosphamide — Cyclophosphamide (750mg/m2/day x 2 days Intravenous (IV)) is administered as pre-treatment medication of TBI-1301.
Drug: Fludarabine — Fludarabine (30mg/m2/day x 2 days Intravenous (IV)) is administered as pre-treatment medication of TBI-1301.

SUMMARY:
The purpose of this study is to verify the safety and the efficacy of TBI-1301 for NY-ESO-1 expressing synovial sarcoma when administered following cyclophosphamide/fludarabine pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Histologically confirmed synovial sarcoma
3. Surgically unresectable tumor
4. Progressing or recurrent synovial sarcoma which has been treated with 1-4 regimens of systemic chemotherapies including anthracycline
5. HLA-A*02:01 or HLA-A*02:06 positive
6. Tumor that express NY-ESO-1 by immunohistochemistry
7. Measurable lesions that are evaluable by the RECIST ver1.1
8. ECOG Performance Status of 0, 1 or 2
9. No treatment such as chemotherapy and be expected to recover fully from the previous treatment at the time of the lymphocytes collection for manufacturing
10. Life expectancy ≥ 16 weeks after consent
11. No severe damage on the major organs (bone marrow, heart, lung, liver, kidney, etc) and meet the following lab value criteria; Total bilirubin ≤ 1.5 x upper limit of normal (ULN); AST(GOT), ALT(GPT) < 3.0 x ULN; Creatinine < 1.5 x ULN; 2,500/μL < WBC ≤ULN; Hemoglobin ≥ 8.0g/dL; Platelets ≥ 75,000/μL
12. Patients must be able to understand the study contents and to give a written consent at his/her free will.

Exclusion Criteria:

1. Patients with the following conditions are excluded from the study; Unstable angina, cardiac infarction, or heart failure; Uncontrolled diabetes or hypertension; Active infection; Obvious interstitial pneumonia or lung fibrosis by chest X-ray; Active autoimmune disease requiring steroids or immunosuppressive therapy.
2. Active metastatic tumor cell invasion into CNS
3. Active multiple cancer
4. Positive for HBs antigen or HBV-DNA observed in serum
5. Positive for HCV antibody and HCV-RNA observed in serum
6. Positive for antibodies against HIV or HTLV-1
7. History of serious hypersensitivity reactions to bovine or murine derived substances.
8. History of hypersensitivity reaction to ingredients or excipients of investigational drugs used in this study
9. History of hypersensitivity reaction to antibiotics used in manufacturing for the investigational drug used in this study.
10. History of treatment with cell therapy or gene therapy
11. Alcohol or drug dependence that may interfere with study participation
12. Pregnant females, lactating females (except when they cease and do not resume lactation) or female and male patients who cannot agree to practice the adequate birth control from the consent to 6 months after infusion of the investigational drug.
13. Clinically significant systemic illness that in the judgment of the PI or sub-investigator would compromise the patient's ability to tolerate protocol therapy or significantly increase the risk of complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 52 weeks
  Evaluate response rate by measuring response using RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Kyusyu University Hospital, Fukuoka, Japan